CLINICAL TRIAL: NCT06277713
Title: Preventing Exercise Resistance With Sedentary Interruptions
Acronym: PERSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Principal investigator, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CME2023/069
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Sedentary Behavior; Lipid Metabolism Disorder; Exercise
Keywords: Exercise; Postprandial metabolism
MeSH Terms: conditions — Sedentary Behavior; Lipid Metabolism Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will follow three regimes of 2 days each including a sedentary control, a sedentary with exercise and a standing breaks with exercise regimen. The sequence of the regimens will be randomised. Each regimen will be followed by a minimum wash-out period of 7 days during which subjects will continue their normal lifestyle.
  We will use a balanced design with 6 randomisation blocks (ABC, ACB, BAC,BCA, CAB, CBA). The randomisation will be computer-generated and allocation will be determined by a member of the research team drawing a sealed, non-translucent envelop with herein written the scheme.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the allocation of participants as samples will be code labeled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise after prolonged sitting (SIT) (Active Comparator): All participants will be instructed to complete two working days (8h) where they perform seated desk-work throughout the day. At the end of the second day, they will perform a supervised exercise bout at the research facility.
  Interventions: Behavioral: Exercise bout; Behavioral: Sedentary
- Exercise after sitting with standing breaks (WBR) (Experimental): All participants will be instructed to complete two working days (8h) where they alternate seated desk-work with standing desk-work hourly throughout the day. At the end of the second day, they will perform a supervised exercise bout at the research facility.
  Interventions: Behavioral: Standing interruptions; Behavioral: Exercise bout
- Non-exercise control (NEX) (Other): In this control group all participants will be instructed to complete two working days (8h) where they perform seated desk-work throughout the day.
  Interventions: Behavioral: Sedentary

INTERVENTIONS:
Behavioral: Standing interruptions — A mobile sit-to-stand desk will be installed at the workplace and participants are instructed to alternate their working position every 30 minutes during two working days (8h).
  Arms: Exercise after sitting with standing breaks (WBR)
Behavioral: Exercise bout — Participants will perform a continuous aerobic exercise bout for a duration of 60 minutes at a moderate intensity, which is defined as 60% of their maximal oxygen uptake (VO2max).
  Arms: Exercise after prolonged sitting (SIT); Exercise after sitting with standing breaks (WBR)
Behavioral: Sedentary — Participants are instructed to minimise any behaviour that is not sedentary during two working days (8h).
  Arms: Exercise after prolonged sitting (SIT); Non-exercise control (NEX)

SUMMARY:
The goal of this randomised cross-over trial is to learn about the interaction between sedentary behaviour throughout the day and the metabolic effect of an exercise bout on that same day in office workers with an increased risk for chronic disease.

The main question this study aims to answer is if the lipid-lowering effects of an exercise bout can be more pronounced by implementing alternations between a seated and a standing working position throughout the day.

Participants will be asked to:

* Complete three intervention periods for a duration of 2 days at their workplace,
* Attend a supervised training session (60min) at the research facility at the end of each intervention period,
* Attend three assessment days at the research facility where postprandial metabolism will be evaluated after a standardised meal test.

DETAILED DESCRIPTION:
The World Health Organisation recently published guidelines with physical activity recommendations that serve to promote healthy lifestyles and thus can help reduce the risk of chronic diseases. In these, they also included for the first time that sedentary behaviour (e.g. sedentary work, driving a car, ...) should be reduced as much as possible since there are clear links between a sedentary lifestyle and negative health effects.

However, WHO also indicates that more research is needed to investigate the health effects of interactions between planned physical activity and sedentary behaviour. This is of even greater importance as there are now some studies indicating that the acute effects of an exercise session are greatly reduced when combined with prolonged sitting throughout the day. This new insight has been labelled as sitting-induced exercise resistance. This study aims to investigate whether it is possible to reduce sitting behaviour by moving more and optimally preserve the effects of a training session.

This study will evaluate how the combination of sitting behaviour and a training session affects certain health parameters. Indeed, prolonged sitting leads to an increased risk of poor cardiometabolic health and consequently an increased risk of developing conditions such as diabetes and cardiovascular disease. Recent research shows that interrupting prolonged sitting can largely prevent some adverse effects on cardiometabolic health. Furthermore, it also shows that the positive effects of an exercise session are greatly reduced when this workout is scheduled on a day that was otherwise spent mainly sitting.

Previous research shows that interrupting sitting behaviour after 20 minutes by short-term (2min) exercise at light intensity would be optimal to improve glucose metabolism. However, this pattern is not very practical to apply in a work environment. For this, installing sit-stand desks could be a solution, as it seems that introducing such sit-stand desks in a work environment could cost-effectively reduce the risk of developing a number of chronic diseases by reducing sitting time. In this study, the effects on postprandial lipemia of reducing prolonged sitting time by introducing sit-stand desks and an exercise bout will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* between 30 and 65 years old,
* primarily work in an office environment for at least 0.75 full time equivalents,
* sedentary (on average >9h of sedentary time per day, assessed objectively),
* at an increased risk for disturbances in lipid profile (assessed with fingerstick (Analox®) total cholesterol >200 mg/dL or fingerstick triglycerides >150 mg/dL),
* written informed consent to participate in the study.

Exclusion Criteria:

* medical conditions precluding physical activity (PA) participation,
* abusive alcohol intake (>20 units/week),
* pregnant or intention to become pregnant,
* change in dietary habits or weight loss (>2kg) in the last month before the study,
* a diagnosis of cardiometabolic diseases such as diabetes mellitus or cardiovascular diseases.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Total and incremental area under the curve of postprandial response in lipid metabolism | 360 minutes
  Lipid levels will be assessed at nine different timepoints (0 minutes, 30 minutes, 60 minutes, 120 minutes, 180 minutes, 210 minutes, 240 minutes, 300 minutes and 360 minutes). Postprandial responses will be defined as the area under the curve (AUC) over the three-hour period after each test meal and the cumulative AUC of the whole time frame.

SECONDARY OUTCOMES:
Total and incremental area under the curve of glucose and insulin postprandial responses | 360 minutes
  Glucose and insulin levels will be assessed at nine different timepoints (0 minutes, 30 minutes, 60 minutes, 120 minutes, 180 minutes, 210 minutes, 240 minutes, 300 minutes and 360 minutes). Postprandial responses will be defined as the area under the curve (AUC) over the three-hour period after each test meal and the cumulative AUC of the whole time frame.
Resting metabolic rate | 0 minute
  Resting metabolic rate will be determined by indirect calorimetry on the morning of each assessment day.

CONTACTS AND LOCATIONS:
Overall Officials: Bert Op 't Eijnde, Prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Yes
In a restriced access depositry. Personal data is sensitive data and is thus protected in a restricted access repository. During the project these data will be pseudonymized and after completion of the project data will be anonymized and the pseudonymization key will be destroyed. Access can be granted by the primary investigator who holds the pseudonymization key in a restricted folder during the project.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the results, data will become available for a duration of 25 years.
Access Criteria: Access will be granted after motivated and reasonable request to the principal investigator.